CLINICAL TRIAL: NCT02825472
Title: Exercise Training in Grown-up Congenital Heart Disease
Acronym: ExTra-GUCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Berto J Bouma, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL5378201815
Record Dates: First submitted 2016-06-23; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease; Sport; Exercise training
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise training program (Active Comparator): Six-months sports participation, three times per week for 30 minutes in the target heart rate zone
  Interventions: Behavioral: exercise training
- No exercise training program (No Intervention): no exercise training program, usual care

INTERVENTIONS:
Behavioral: exercise training — 3 times per week 30 minutes of exercise training in the target heart rate zone
  Arms: Exercise training program

SUMMARY:
Rationale: Regular physical activity and aerobic exercise training are related to decreased cardiovascular mortality in healthy individuals, as well as in individuals with cardiovascular risk factors and cardiac patients. Unfortunately, no such data is available on exercise training in adult patients with congenital heart disease.

Objective: The objective of the ExTra GUCH trial is to assess whether encouragement of a six-month sports participation program in addition to usual care in symptomatic adult patients with congenital heart disease improves exercise capacity and quality of life, and lowers serum N-terminal prohormone brain natriuretic peptide (NT-proBNP) levels.

Study design: International, multi-centre parallel randomized controlled trial.

Study population: Adult patients with congenital heart disease, who are in New York Heart Association (NYHA) class II or III.

Intervention (if applicable): The intervention group receives a six-month individualized exercise training program, the control group receives usual care.

Main study parameters/endpoints: The primary outcome is the change in peakVO2 between patients in the sports participation group, and the control group. Secondary outcome measures are change in NYHA functional class, quality of life, and NT-proBNP levels. The primary safety outcome is the composite of all hospitalizations, and all deaths during, or within three hours after exercise. The secondary safety outcome is the composite of all exercise related injuries for which medical attention is sought.

DETAILED DESCRIPTION:
The investigators intend to submit the trial design of this study for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Congenital heart disease of all complexities
* NYHA Class II or III

Exclusion Criteria:

* Inability to give informed consent
* Inability to participate in an exercise training program
* Exercise-induced arrhythmia and/or ischemia
* Cyanosis at rest
* Pregnancy
* Major cardiovascular event and/or procedure within three months previous to inclusion.
* Participation in interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint: change in peak VO2 | 6 months
  change in peak VO2 between baseline and 6-months follow-up CPET
Primary safety endpoint: composite of hospitalizations, deaths during, or within three hours after exercise | between 3 hours after exercise for the duration of the 6 months study period
  The primary safety outcome is the composite of all hospitalizations, and all deaths during, or within three hours after exercise.

SECONDARY OUTCOMES:
Secondary efficacy endpoint: quality of life | 6 months
  change in SF36 scores between baseline and 6-months follow-up
Secondary efficacy endpoint: NTproBNP level | 6 months
  change in NTproBNP between baseline and 6-months follow-up
Secondary safety endpoint: composite of all exercise related injuries for which medical attention is sought | 6 months study period
  The secondary safety outcome is the composite of all exercise related injuries for which medical attention is sought during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Mulder, MD, PhD, Principal Investigator — AIDS Malignancy Consortium
Locations (2):
- Department of Cardiology, I.R.C.C.S. Policlinico San Donato Milanese, Milan, Piazza Edmondo Malan, Italy
- Hospital, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No